CLINICAL TRIAL: NCT00783315
Title: Practice-Based Opportunities for Weight Reduction Trial at Johns Hopkins
Brief Title: Evaluating Weight Loss Programs for Obese People at Risk for Heart Disease (The POWER Study)
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Healthways, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00012877; U01HL087085 (NIH)
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Hypertension; Diabetes; Hypercholesterolemia
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus; Hypercholesterolemia | interventions — Weight Reduction Programs

STUDY DESIGN:
Intervention Model Description: Three Group:
  1. advice only comparison group
  2. remotely delivered behavioral weight loss group
  3. in-person behavioral weight loss group
Who Masked: Outcomes Assessor
Masking Description: Persons who measured weight and other outcomes were masked to randomized assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Self-Directed Weight Loss Program (Control Group)
  Interventions: Behavioral: Self-Directed Weight Loss Program
- 2 (Experimental): Call-Center Directed (CCD) Weight Loss Program
  Interventions: Behavioral: Call-Center Directed (CCD) Weight Loss Program
- 3 (Experimental): In-Person Directed (IPD) Weight Loss Program
  Interventions: Behavioral: In-Person Directed (IPD) Weight Loss Program

INTERVENTIONS:
Behavioral: Call-Center Directed (CCD) Weight Loss Program — This program will be implemented by trained counselors of Healthways, Inc., and will use telephone, Web, and e-mail contacts to engage participants. There will be no in-person visits.
  Arms: 2
Behavioral: In-Person Directed (IPD) Weight Loss Program — This program will be primarily implemented through in-person visits (including group sessions) with health counselors at Johns Hopkins University. Telephone, Web, and e-mail contacts will occasionally be used.
  Arms: 3
Behavioral: Self-Directed Weight Loss Program — Participants will meet with study staff at the beginning of the study and will receive written information about weight loss.
  Arms: 1

SUMMARY:
Many people who are obese also have high blood pressure, high cholesterol, or diabetes-all conditions that can increase the risk of heart disease. This study will evaluate two programs that aim to encourage weight loss among obese people who are at risk for developing heart disease.

DETAILED DESCRIPTION:
High blood pressure, high cholesterol, and diabetes are all conditions that increase a person's risk of developing heart disease. Many people with these conditions are also overweight, and it is recommended that such people lose weight to reduce their risk of heart disease. Previous weight loss studies have mainly examined in-person weight loss programs and not Web- or e-mail-based weight loss programs. In addition, the primary care providers of participants in these previous studies typically had no direct involvement in the programs. This study will compare two weight loss programs-an In-Person Directed (IPD) program, which is primarily comprised of in-person visits with health counselors, and a Call-Center Directed (CCD) program, which uses only telephone, Web sites, and e-mail to contact and counsel participants. These two programs will also be compared against a self-directed weight loss program, which will act as a control group. The ultimate purpose of this study is to evaluate the effectiveness of the IPD, CCD, and self-directed programs at increasing weight loss and reducing risk factors in obese people at risk of developing heart disease.

This study will enroll overweight adults who have high blood pressure, high cholesterol, or diabetes. Participants will attend a baseline study visit for weight and blood pressure measurements. They will then be randomly assigned to participate in one of the following three programs for 2 years.

1. IPD Program: This program will be directed by health counselors from Johns Hopkins University. For Months 1 to 3, participants will attend a group or individual meeting with a counselor each week. For Months 4 to 6, meetings will be held three times a month; after Month 6, meetings will occur twice a month. Some of these meetings may be held over the phone or by e-mail. Participants will keep a food and exercise diary and they will enter their weight and calorie consumption on the study Web site. Study researchers will provide participants' doctors with relevant information on participants' weight loss.
2. CCD Program: This program will be directed by counselors from Healthways, Inc., a company that assists individuals in managing their medical problems. All contacts will occur by phone, e-mail, or the Web; there will be no in-person visits. Participants will be able to review weight loss information on the study Web site. For Months 1 to 3, participants will contact their counselors each week. For Months 4 to 6, contact with study counselors will occur at least once a month; after Month 6, contact with study counselors will occur every other month. Participants will keep a food and exercise diary and they will enter their weight and calorie consumption on the study Web site. Study researchers will provide participants' doctors with relevant information on participants' weight loss.
3. Self-Directed Program: In this program, study staff will meet with participants once at the beginning of the study, at which time participants will receive written information about losing weight. Participants will also receive access to a study Web site that has information about weight loss.

All participants will attend study visits at Months 6, 12, and 24 and at the end of the study, which is anticipated to be in February 2011. Study researchers will also collect information by phone at Month 18. At each study visit, participants will complete questionnaires; provide blood samples; and undergo measurements of weight, waist, and blood pressure. A portion of blood may be stored for future studies; this will be optional.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension, hypercholesterolemia, and/or diabetes mellitus, all of which are treated with medication, measured in the clinic, or confirmed by primary care provider (systolic blood pressure greater than or equal to 140 mm Hg, diastolic blood pressure greater than or equal to 90 mm Hg, low density lipoprotein cholesterol [LDL-C] greater than or equal to 130 mg/dL, or fasting blood sugar greater than 125 mg/dL)
* BMI of at least 30 to 50 kg/m2 and weight less than or equal to 400 lbs
* Willing to change diet, physical activity, and weight
* Willing to be randomly assigned to any of the study groups
* Patient of a participating doctor
* Patient self-reports two doctor visits in the 12 months before study entry
* Demonstrated use of Web and e-mail
* Access to Internet at least 4 days per week
* People with the following conditions are eligible to enroll in the study with primary care provider approval:

  1. Diabetes mellitus
  2. Prior cardiovascular disease event more than 6 months before study entry
  3. Known stable cardiovascular disease or peripheral vascular disease
  4. Screen positive on Rose Questionnaire

Exclusion Criteria:

* Heart attack, stroke, or atherosclerotic cardiovascular disease (ASCVD) procedure in the 6 months before study entry
* Serious medical condition that is likely to hinder accurate measurement of weight, for which weight loss is not advisable, or that would cause weight loss [e.g., end-stage renal disease (ESRD) on dialysis, cancer diagnosis or treatment in the 2 years before study entry]
* Prior or planned bariatric surgery
* Use of prescription weight loss medication, including off-label drugs (e.g., topiramate, bupropion, byetta) or over-the-counter orlistat in the 6 months before study entry
* Long-term use (in the 6 months before study entry) of medications likely to cause weight gain or prevent weight loss (e.g., corticosteroids, lithium, olanzapine, risperidone, clozapine)
* Unintentional weight loss in the 6 months before study entry (greater than or equal to 5% of body weight)
* Intentional weight loss in the 6 months before study entry (greater than or equal to 5% of body weight)
* Pregnant or breastfeeding in the 6 months before study entry
* Planning to become pregnant in the 2 years after study entry
* Planning to relocate from area in the 2 years after study entry
* Another member of the household is a study participant or study staff member
* Self-reported average consumption of more than 14 alcoholic drinks each week
* Psychiatric hospitalization in the 1 year before study entry
* Unstable angina
* Blood pressure greater than 160/100 mm Hg

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2011-02-28 (Actual); Study Completion 2011-02-28 (Actual)

PRIMARY OUTCOMES:
Weight | Measured at Month 24

SECONDARY OUTCOMES:
Blood pressure | Measured at Month 24
Hypertension control | Measured at Month 24
Homeostasis model assessment of insulin resistance (HOMA-IR) | Measured at Month 24
Framingham risk | Measured at Month 24
Metabolic syndrome | Measured at Month 24
Body mass index (BMI) | Measured at Month 24
Lipid levels | Measured at Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J. Appel, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- ProHealth, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bennett WL, Wang NY, Gudzune KA, Dalcin AT, Bleich SN, Appel LJ, Clark JM. Satisfaction with primary care provider involvement is associated with greater weight loss: Results from the practice-based POWER trial. Patient Educ Couns. 2015 Sep;98(9):1099-105. doi: 10.1016/j.pec.2015.05.006. Epub 2015 May 27. PMID 26026649
- [Derived] Jerome GJ, Dalcin A, Coughlin JW, Fitzpatrick S, Wang NY, Durkin N, Yeh HC, Charleston J, Pozefsky T, Daumit GL, Clark JM, Louis TA, Appel LJ. Longitudinal accuracy of web-based self-reported weights: results from the Hopkins POWER Trial. J Med Internet Res. 2014 Jul 15;16(7):e173. doi: 10.2196/jmir.3332. PMID 25042773
- [Derived] Bennett WL, Gudzune KA, Appel LJ, Clark JM. Insights from the POWER practice-based weight loss trial: a focus group study on the PCP's role in weight management. J Gen Intern Med. 2014 Jan;29(1):50-8. doi: 10.1007/s11606-013-2562-6. Epub 2013 Sep 4. PMID 24002616
- [Derived] Appel LJ, Clark JM, Yeh HC, Wang NY, Coughlin JW, Daumit G, Miller ER 3rd, Dalcin A, Jerome GJ, Geller S, Noronha G, Pozefsky T, Charleston J, Reynolds JB, Durkin N, Rubin RR, Louis TA, Brancati FL. Comparative effectiveness of weight-loss interventions in clinical practice. N Engl J Med. 2011 Nov 24;365(21):1959-68. doi: 10.1056/NEJMoa1108660. Epub 2011 Nov 15. PMID 22085317
- [Derived] Yeh HC, Clark JM, Emmons KE, Moore RH, Bennett GG, Warner ET, Sarwer DB, Jerome GJ, Miller ER, Volger S, Louis TA, Wells B, Wadden TA, Colditz GA, Appel LJ. Independent but coordinated trials: insights from the practice-based Opportunities for Weight Reduction Trials Collaborative Research Group. Clin Trials. 2010 Aug;7(4):322-32. doi: 10.1177/1740774510374213. Epub 2010 Jun 23. PMID 20573639